CLINICAL TRIAL: NCT05115890
Title: Mechanisms of Impaired Skeletal Muscle Blood Flow and Exercise Intolerance in Veterans With Heart Failure With Preserved Ejection Fraction: Efficacy of Knee Extensor Training
Brief Title: Muscle Blood Flow Regulation in HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: F3670-W
Record Dates: First submitted 2021-10-21; First posted 2021-11-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: HFpEF
Keywords: HFpEF; Muscle Blood Flow; Exercise Tolerance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients with HFpEF assigned to 8 weeks of exercise training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise training (Experimental): Patients with HFpEF will participate in the 8 weeks of supervised, two-legged, knee extensor exercise training for 3 days per week. Each exercise session will involve a 5-min warm-up and a 5-min cool-down, and exercise intensity will range between 40%-90% of maximal work rate. Maximal work rate will be re-assessed every two weeks.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Patients with HFpEF will undergo 8 weeks of exercise training.

SUMMARY:
Heart failure with preserved ejection (HFpEF) disproportionately affects Veterans and is the number one reason for hospital discharge in the VA Health Care System. Exercise intolerance is a common complication experienced by patients with HFpEF, perpetuating physical inactivity and accelerating disease progression. This research proposal aims to elucidate mechanisms responsible for inadequate skeletal muscle blood flow and exercise intolerance in patients with HFpEF compared with healthy controls as well as following 8 weeks of exercise training in patients with HFpEF only.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF) disproportionately afflicts Veterans and is the leading cause of hospitalization and mortality within the VA Health Care System. One chief symptom of HFpEF is severe exercise intolerance, an important predictor of quality of life, functional capacity, and mortality. In these patients, severe exercise intolerance is attributable to a disease-related loss of "peripheral vascular control," as evidenced by a marked attenuation in exercising skeletal muscle blood flow. Loss of peripheral vascular control is manifested as dysfunctions of the autonomic nervous system (ANS) and vasodilatory ability of the microvasculature, thereby restraining skeletal muscle blood flow and O2 delivery and limiting the capacity for sustained physical activity. This research proposal aims to elucidate peripheral vascular control mechanisms responsible for inadequate skeletal muscle blood flow and exercise intolerance in patients with HFpEF. In addition, there is some indication that aerobic exercise training may improve peripheral vascular function in HFpEF , though the mechanisms have yet to be elucidated. Thus, an additional aim of this research proposal is to evaluate peripheral vascular control mechanisms of skeletal muscle blood flow and exercise tolerance following 8 weeks of exercise training in patients with HFpEF. To test this, the initial phase will involve a cross-sectional comparison of patients with HFpEF (n=35) and age and sex-matched healthy controls (n=35), followed by an interventional phase where only patients with HFpEF will enter 8 weeks of exercise training. It is anticipated that knowledge gained will (a) improve the understanding of HFpEF pathophysiology and (b) determine the efficacy of a unique exercise training modality to restore functional capacity and exercise tolerance in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and able to give written informed consent
* New York Heart Association (NYHA) functional class II or III
* Left Ventricular Ejection Fraction (LVEF) > 50%
* Plasma Brain Natriuretic Peptide (BNP) >200 pg/mL or NT-proBNP 400 pg/mL at enrollment

Exclusion Criteria:

* Prior EF of <50%.
* NYHA Class IV or HF that cannot be stabilized on optimized pharmacotherapy
* Acute coronary syndrome, infiltrative cardiomyopathy, or myocarditis
* Patients with HFpEF secondary to significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction)
* Orthopedic limitations that would prohibit knee-extensor exercise
* Women currently taking hormone replacement therapy (HRT) will be excluded from the proposed studies due to the direct vascular effects of HRT
* Women who are pregnant or may become pregnant, but the typical age of female patients with HFpEF will be postmenopausal
* Current smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | Change from baseline six-minute walk test distance at 8 weeks
  The six-minute walk test is used to measure distance covered during walking at a comfortable speed for six minutes
Muscle blood flow | Change from baseline skeletal muscle blood flow at 8 weeks
  Muscle blood flow will be assessed non-invasively via Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Kanokwan Bunsawat, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No